CLINICAL TRIAL: NCT02292784
Title: Follow-Up Study to Assess Long-Term Safety and Outcomes in Infants and Children Born to Mothers Participating in Retosiban Treatment Studies
Brief Title: Follow up Study to Assess Long Term Safety and Outcomes in Infants and Children Born to Mothers Participating in Retosiban Treatment Studies
Acronym: ARIOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 200722
Record Dates: First submitted 2014-11-13; First posted 2014-11-17 (Estimated); Results first posted 2020-07-09 (Actual); Last update posted 2020-07-09 (Actual); Status verified 2020-06

CONDITIONS: Obstetric Labour, Premature
Keywords: infants; retosiban; Preterm Labor; long-term safety follow-up
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature | interventions — GSK221149A; atosiban

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (200719 study) (Placebo Comparator): All infants and children born to women who received the placebo (0.9 percent sodium chloride infusion matched for retosiban volume, intravenous [IV] loading dose over 5 minutes and continuous infusion rate including dose increase in participants with an inadequate response any time after first hour of treatment) in 200719 study. Current study will not require any medical interventions or study visits to an investigational site.
  Interventions: Drug: Placebo
- Retosiban (200719 and 200721 study) (Experimental): All infants and children born to women who received retosiban (6 milligram [mg] IV loading dose of retosiban over 5 minutes followed by a 6 mg per hour continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg per hour continuous infusion for remainder of 48-hour treatment period) in 200719 study or 200721 study. Current study will not require any medical interventions or study visits to an investigational site.
  Interventions: Drug: Retosiban
- Atosiban (200721 study) (Active Comparator): All infants and children born to women who received atosiban (in 3 successive stages; an initial bolus dose of 6.75 mg using atosiban 6.75 mg per 0.9 milliliter [mL] solution for injection, followed by continuous high dose infusion at 18 mg per hour for 3 hours, then a lower 6 mg per hour infusion for the remainder of the 48-hour using the atosiban 37.5 mg per 5 mL concentrate for solution) in 200721 study. Current study will not require any medical interventions or study visits to an investigational site.
  Interventions: Drug: Atosiban

INTERVENTIONS:
Drug: Retosiban — This is a safety follow-up study of infants and children exposed to retosiban during their mother's participation in a Phase III treatment study for SPTL. Infants enrolled in this study will not be administered any investigational product.
  Arms: Retosiban (200719 and 200721 study)
Drug: Atosiban — This is a safety follow-up study of infants and children exposed to atosiban comparator during their mother's participation in a Phase III treatment study for SPTL. Infants enrolled in this study will not be administered any investigational product.
  Arms: Atosiban (200721 study)
Drug: Placebo — This is a safety follow-up study of infants and children exposed to matching placebo for retosiban/ atosiban during their mother's participation in a Phase III treatment study for SPTL. Infants enrolled in this study will not be administered any investigational product
  Arms: Placebo (200719 study)

SUMMARY:
The primary objective of this study is to assess the safety and outcomes of infants and children who were exposed to retosiban or comparator in utero in the Phase III spontaneous preterm labor (SPTL) treatment studies, to provide assurance that treatment is not associated with significant adverse outcomes in early childhood. The enrolled infants and children will be followed at pre-specified intervals until they reach 24 months chronological age. This study does not require medical interventions or study visits to an investigational site, instead, parents or legal guardians will be prompted at certain time points to complete developmental questionnaires and other data on their children's health status via an electronic device. Data collected during the infant and child follow up study will be managed by a centralized research coordinating center (RCC). Regionally based pediatricians will serve as study principal investigators (referred to as RCC-PIs) for this study. All communications the RCC-PI has with the parent/legal guardian or the child's health care provider (HCP) will occur remotely; there will be no clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* Mother is randomly assigned and dosed (retosiban or comparator) in 1 of the Phase III SPTL retosiban clinical studies.
* Infant is alive at 28 days post EDD.
* Written informed consent is obtained from the parent(s) or legal guardian(s) of the infant. The parent/legal guardian of subjects aged 12 to 17 years must also provide written agreement for the infant to participate in the study where required by applicable regulatory and country or state requirements.

Exclusion Criteria:

* There are no formal exclusion criteria for participation.

Ages: 10 Weeks to 20 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 98 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-09-02 (Actual); Study Completion 2019-09-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (25):
- United States (2):
  - GSK Investigational Site, Park Ridge, Illinois
  - GSK Investigational Site, Galveston, Texas
- GSK Investigational Site, Ghent, Belgium
- Germany (2):
  - GSK Investigational Site, Freiburg im Breisgau, Baden-Wurttemberg
  - GSK Investigational Site, Jena
- Israel (7):
  - GSK Investigational Site, Hadera
  - GSK Investigational Site, Haifa
  - GSK Investigational Site, Holon
  - GSK Investigational Site, Kfar Saba
  - GSK Investigational Site, Petah Tikva
  - GSK Investigational Site, Safed
  - GSK Investigational Site, Tel Aviv
- Italy (2):
  - GSK Investigational Site, Siena, Tuscany
  - GSK Investigational Site, Monza
- Japan (2):
  - GSK Investigational Site, Miyagi
  - GSK Investigational Site, Miyazaki
- Mexico (3):
  - GSK Investigational Site, Guadalajara, Jalisco
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Ciudad Obregón, Sonora
- South Korea (2):
  - GSK Investigational Site, Seongnam
  - GSK Investigational Site, Seoul
- GSK Investigational Site, Zaragoza, Spain
- GSK Investigational Site, Uppsala, Sweden
- United Kingdom (2):
  - GSK Investigational Site, Sunderland, Tyne & Wear
  - GSK Investigational Site, London

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Powell M, Saade GR, Thornton S, Pimenta JM, Haque N, Miller D, Beach KJ, Snidow J, Correa EO, Scott R. Safety and Outcomes in Infants Born to Mothers Participating in Retosiban Treatment Trials: ARIOS Follow-up Study. Am J Perinatol. 2023 Jul;40(10):1135-1148. doi: 10.1055/s-0041-1733784. Epub 2021 Aug 5. PMID 34352924

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomized, long-term follow-up study to evaluate the safety and outcomes of infants and children born to women who received retosiban or comparator in the Phase III spontaneous preterm labor (SPTL) treatment studies:200719 (NCT02377466) and 200721 (NCT02292771). Current study was referred as a retosiban infant outcome study (ARIOS).
Pre-assignment Details: A total of 101 participants were screened and 98 participants were enrolled and randomized in this study.
Groups:
- Placebo (200719 Study): All infants and children born to women who received the placebo (0.9 percent sodium chloride infusion matched for retosiban volume, intravenous [IV] loading dose over 5 minutes and continuous infusion rate including dose increase in participants with an inadequate response any time after first hour of treatment) in 200719 study. Current study did not require any medical interventions or study visits to an investigational site.
- Atosiban (200721 Study): All infants and children born to women who received atosiban (in 3 successive stages; an initial bolus dose of 6.75 milligram [mg] using atosiban 6.75 mg per 0.9 milliliter [mL] solution for injection, followed by continuous high dose infusion at 18 mg per hour for 3 hours, then a lower 6 mg per hour infusion for the remainder of the 48-hour using the atosiban 37.5 mg per 5 mL concentrate for solution) in 200721 study. Current study did not require any medical interventions or study visits to an investigational site.
- Retosiban (200719 and 200721 Study): All infants and children born to women who received retosiban (6 mg IV loading dose of retosiban over 5 minutes followed by a 6 mg per hour continuous infusion of retosiban over 48 hours. Participants with an inadequate response any time after first hour of treatment were administered another 6 mg retosiban loading dose followed by 12 mg per hour continuous infusion for remainder of 48-hour treatment period) in 200719 study or 200721 study. Current study did not require any medical interventions or study visits to an investigational site.
Period: Overall Study
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Started | 5 | 44 | 49
Completed | 4 | 24 | 28
Not Completed | 1 | 20 | 21
Not completed — Lost to Follow-up | 1 | 17 | 18
Not completed — Withdrawal by Subject | 0 | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study) | Total
Number analyzed (Participants) | 5 | 44 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: Months] | 2.16 (1.479) | 2.18 (1.158) | 2.12 (0.932) | 2.15 (1.056)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 18 | 21 | 40
  Male | 4 | 26 | 28 | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/African (Afr) Heritage | 0 | 1 | 1 | 2
  American Indian or Alaskan Native | 0 | 5 | 6 | 11
  Asian-Central/South Asian Heritage | 0 | 0 | 1 | 1
  Asian-East Asian Heritage | 1 | 4 | 8 | 13
  Asian-Japanese Heritage | 4 | 0 | 2 | 6
  White-Arabic/North Afr/Caucasian/European Heritage | 0 | 34 | 31 | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants and Children With Newly Diagnosed Chronic Medical Conditions (After 28 Days Post Estimated Date of Delivery)
Description: The parents of the infants filled in an online child health inventory (CHI) questionnaire, which asked them about each condition. If they reported anything, it was then verified by a healthcare professional. Number of infants and children with newly diagnosed chronic medical conditions are presented.
Time Frame: From 28 days post estimated date of delivery up to 24 months
Population: ARIOS Safety Population was a subset of the Infant Safety Population (all the infants whose mothers were randomized and received retosiban or comparator in any of the Phase III treatment trials) for which the mother/infant pairs were enrolled into the ARIOS study.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants | 0 | 1 | 3

2. Primary Outcome: Number of Infants and Children With Newly Diagnosed Congenital Anomalies (After 28 Days Post Estimated Date of Delivery)
Description: A congenital anomaly is a condition present at birth that results from malformation, deformation, or disruption in 1 or more parts of the body, a chromosomal abnormality, or a known clinical syndrome. Congenital anomaly serious adverse events (SAEs) were examined by the birth defect evaluator. Events were coded per centers for disease control and prevention (CDC) Metropolitan Atlanta congenital defects program (MACDP) criteria and/or European surveillance of congenital anomalies (EUROCAT) criteria. Predefined defect codes specified whether the defect was face and neck, a cleft lip or palate, cardiovascular, respiratory, upper gastrointestinal, female genitalia, male genitalia, renal and urinary system, other musculoskeletal defects, skin, a chromosome anomaly, other organ systems, or a specified syndrome. Number of infants and children with newly diagnosed congenital anomalies reported up to 1 year of chronological age and reported after 1 year of chronological age are presented.
Time Frame: From 28 days post estimated date of delivery up to 24 months
Population: ARIOS Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  Up to 1 year of chronological age | 0 | 0 | 2
  After 1 year of chronological age | 0 | 0 | 0

3. Primary Outcome: Number of Infant and Child Death (After 28 Days Post Estimated Date of Delivery)
Description: Number of infant and child death that occurred after 28 days post estimated date of delivery and up to 24 months are presented.
Time Frame: From 28 days post estimated date of delivery up to 24 months
Population: ARIOS Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Any Domain at 9 Months
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for communication was 13.97, gross motor was 17.82, fine motor was 31.32, problem solving was 28.72 and personal social skills was 18.91. Total score was derived by taking mean of all 5 components. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for any domains in the black zone at 9 months is presented.
Time Frame: At 9 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 3 | 17 | 20
Participants | 0 | 4 | 4

5. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Any Domain at 18 Months
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 18 months, the pre-defined cut-off score for communication was 13.06, gross motor was 37.38, fine motor was 34.32, problem solving was 25.74 and personal social skills was 27.19. Total score was derived by taking mean of all 5 components. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for any domains in the black zone at 18 months is presented.
Time Frame: At 18 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 3 | 19 | 18
Participants | 2 | 5 | 0

6. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Any Domain at 24 Months
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 24 months, the pre-defined cut-off score for communication was 25.17, gross motor was 38.07, fine motor was 35.16, problem solving was 29.78 and personal social skills was 31.54. Total score was derived by taking mean of all 5 components. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for any domains in the black zone at 24 months is presented.
Time Frame: At 24 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 2 | 19 | 25
Participants | 1 | 2 | 2

7. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Gross Motor Skills
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for gross motor skills was 17.82. At 18 months, the pre-defined cut-off score for gross motor skills was 37.38. At 24 months, the pre-defined cut-off score for gross motor skills was 38.07. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for gross motor skills in the black zone at 9, 18 and 24 months is presented.
Time Frame: 9, 18 and 24 months
Population: ARIOS Safety Population. All 98 participants in the study were included in the analysis (5, 44 and 49 Participants), but only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  9 months, n=3,17,20: number analyzed (Participants) | 3 | 17 | 20
  9 months, n=3,17,20 | 0 | 1 | 0
  18 months, n=3,19,18: number analyzed (Participants) | 3 | 19 | 18
  18 months, n=3,19,18 | 1 | 1 | 0
  24 months, n=2,19,25: number analyzed (Participants) | 2 | 19 | 25
  24 months, n=2,19,25 | 0 | 1 | 0

8. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Fine Motor Skills
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for fine motor skills was 31.32. At 18 months, the pre-defined cut-off score for fine motor skills was 34.32. At 24 months, the pre-defined cut-off score for fine motor skills was 35.16. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for fine motor skills in the black zone at 9, 18 and 24 months is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  9 months, n=3,17,20: number analyzed (Participants) | 3 | 17 | 20
  9 months, n=3,17,20 | 0 | 0 | 2
  18 months, n=3,19,18: number analyzed (Participants) | 3 | 19 | 18
  18 months, n=3,19,18 | 1 | 2 | 0
  24 months, n=2,19,25: number analyzed (Participants) | 2 | 19 | 25
  24 months, n=2,19,25 | 0 | 0 | 0

9. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Communication Skills
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for communication skills was 13.97. At 18 months, the pre-defined cut-off score for communication skills was 13.06. At 24 months, the pre-defined cut-off score for communication skills was 25.17. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for communication skills in the black zone at 9, 18 and 24 months is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  9 months, n=3,17,20: number analyzed (Participants) | 3 | 17 | 20
  9 months, n=3,17,20 | 0 | 1 | 1
  18 months, n=3,19,18: number analyzed (Participants) | 3 | 19 | 18
  18 months, n=3,19,18 | 1 | 0 | 0
  24 months, n=2,19,25: number analyzed (Participants) | 2 | 19 | 25
  24 months, n=2,19,25 | 1 | 1 | 2

10. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Problem Solving Skills
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for problem solving skills was 28.72. At 18 months, the pre-defined cut-off score for problem solving skills was 25.74. At 24 months, the pre-defined cut-off score for problem solving skills was 29.78. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for problem solving skills in the black zone at 9, 18 and 24 months is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  9 months, n=3,17,20: number analyzed (Participants) | 3 | 17 | 20
  9 months, n=3,17,20 | 0 | 1 | 2
  18 months, n=3,19,18: number analyzed (Participants) | 3 | 19 | 18
  18 months, n=3,19,18 | 0 | 1 | 0
  24 months, n=2,19,25: number analyzed (Participants) | 2 | 19 | 25
  24 months, n=2,19,25 | 0 | 1 | 0

11. Primary Outcome: Number of Infants With Ages and Stages Questionnaire-3 (ASQ-3) Score in the Black Zone for Personal Social Skills
Description: The ASQ-3 included 6 questions in each area, designed to assess 5 areas of development: communication skills, gross motor skills, fine motor skills, problem solving skills, and personal social skills. Parents answered either yes (10 points), sometimes (5 points) or not yet (0 points) to each question to complete ASQ-3. At 9 months, the pre-defined cut-off score for personal social skills was 18.91. At 18 months, the pre-defined cut-off score for personal social skills was 27.19. At 24 months, the pre-defined cut-off score for personal social skills was 31.54. Any infant who scored below the cut-off, a score more than or equal to 2 standard deviations below the mean score (that is Black zone in the score chart) in any of the 5 areas of the ASQ-3 was to be referred to a developmental specialist for a formal neurodevelopmental assessment. Number of infants with ASQ-3 scores for personal social skills in the black zone at 9, 18 and 24 months is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 5 | 44 | 49
Participants
  9 months, n=3,17,20: number analyzed (Participants) | 3 | 17 | 20
  9 months, n=3,17,20 | 0 | 2 | 0
  18 months, n=3,19,18: number analyzed (Participants) | 3 | 19 | 18
  18 months, n=3,19,18 | 0 | 1 | 0
  24 months, n=2,19,25: number analyzed (Participants) | 2 | 19 | 25
  24 months, n=2,19,25 | 0 | 1 | 0

12. Primary Outcome: Number of Infants Referred for Developmental Evaluation Using Bayley Scales of Infant Development, Third Edition (BSID-III)
Description: Any infant who scored below the cut-off i.e., a score greater than or equal to 2 Standard Deviations (SDs) below the mean score (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a neurodevelopmental evaluation using the BSID-III. It scaled scores for cognitive, language (receptive and expressive), motor (fine and gross motor). The language and motor areas each have a composite score, with a mean of 100, a SD of 15 and a range of 40 to 160. Scores lower than 70 indicated moderate or severe impairment. In the cognitive area, the infant scored "1" if they could do an activity and "0" if they could not. Total score was derived by taking mean of all the components. Number of infants referred for developmental evaluation using BSID-III is presented.
Time Frame: 9, 18 and 24 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 2 | 5 | 4
Participants
  9 months, n=0,4,4: number analyzed (Participants) | 0 | 4 | 4
  9 months, n=0,4,4 |  | 1 | 3
  18 months, n=2,5,0: number analyzed (Participants) | 2 | 5 | 0
  18 months, n=2,5,0 | 2 | 3 |
  24 months, n=1,2,2: number analyzed (Participants) | 1 | 2 | 2
  24 months, n=1,2,2 | 0 | 2 | 1

13. Primary Outcome: Number of Infants With Bayley Scales of Infant Development, Third Edition Score Greater Than 2 Standard Deviation Below the Mean Score for the Cognitive Scale (Less Than 4)
Description: Any infant who scored below the cut-off i.e., a score greater than or equal to 2 SDs below the mean score (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a neurodevelopmental evaluation using the BSID-III. It scaled scores for cognitive, language (receptive and expressive), motor (fine and gross motor). The language and motor areas each have a composite score, with a mean of 100, a SD of 15 and a range of 40 to 160. Scores lower than 70 indicated moderate or severe impairment. In the cognitive area, the infant scored "1" if they could do an activity and "0" if they could not. Number of infants with BSID-III score greater than 2 SD below the mean score for the cognitive scale (less than 4) is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 0 | 2 | 1
Participants
  9 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  9 months, n=0,0,1 |  |  | 0
  18 months, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  18 months, n=0,2,0 |  | 2 |
  24 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  24 months, n=0,0,1 |  |  | 1

14. Primary Outcome: Number of Infants With Bayley Scales of Infant Development, Third Edition Score Greater Than 2 Standard Deviation Below the Mean Score for the Gross Motor Scale (Less Than 4)
Description: Any infant who scored below the cut-off i.e., a score greater than or equal to 2 SDs below the mean score (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a neurodevelopmental evaluation using the BSID-III. It scaled scores for cognitive, language (receptive and expressive), motor (fine and gross motor). The language and motor areas each have a composite score, with a mean of 100, a SD of 15 and a range of 40 to 160. Scores lower than 70 indicated moderate or severe impairment. In the cognitive area, the infant scored "1" if they could do an activity and "0" if they could not. Number of infants with BSID-III score greater than 2 SD below the mean score for the gross motor scale (less than 4) is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 0 | 2 | 1
Participants
  9 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  9 months, n=0,0,1 |  |  | 0
  18 months, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  18 months, n=0,2,0 |  | 2 |
  24 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  24 months, n=0,0,1 |  |  | 1

15. Primary Outcome: Number of Infants With Bayley Scales of Infant Development, Third Edition Score Greater Than 2 Standard Deviation Below the Mean Score for the Fine Motor Scale (Less Than 4)
Description: Any infant who scored below the cut-off i.e., a score greater than or equal to 2 SDs below the mean score (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a neurodevelopmental evaluation using the BSID-III. It scaled scores for cognitive, language (receptive and expressive), motor (fine and gross motor). The language and motor areas each have a composite score, with a mean of 100, a SD of 15 and a range of 40 to 160. Scores lower than 70 indicated moderate or severe impairment. In the cognitive area, the infant scored "1" if they could do an activity and "0" if they could not. Number of infants with BSID-III score greater than 2 SD below the mean score for the fine motor scale (less than 4) is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 0 | 2 | 1
Participants
  9 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  9 months, n=0,0,1 |  |  | 0
  18 months, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  18 months, n=0,2,0 |  | 2 |
  24 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  24 months, n=0,0,1 |  |  | 1

16. Primary Outcome: Number of Infants With Bayley Scales of Infant Development, Third Edition Score Greater Than 2 Standard Deviation Below the Mean Score for the Language Scale (Less Than 70)
Description: Any infant who scored below the cut-off i.e., a score greater than or equal to 2 SDs below the mean score (i.e., black zone in the score chart) in any of the 5 domains of the ASQ-3 was referred to a developmental specialist for a neurodevelopmental evaluation using the BSID-III. It scaled scores for cognitive, language (receptive and expressive), motor (fine and gross motor). The language and motor areas each have a composite score, with a mean of 100, a SD of 15 and a range of 40 to 160. Scores lower than 70 indicated moderate or severe impairment. In the cognitive area, the infant scored "1" if they could do an activity and "0" if they could not. Number of infants with BSID-III score greater than 2 SD below the mean score for the language scale (less than 70) is presented.
Time Frame: 9, 18 and 24 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 0 | 2 | 1
Participants
  9 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  9 months, n=0,0,1 |  |  | 0
  18 months, n=0,2,0: number analyzed (Participants) | 0 | 2 | 0
  18 months, n=0,2,0 |  | 2 |
  24 months, n=0,0,1: number analyzed (Participants) | 0 | 0 | 1
  24 months, n=0,0,1 |  |  | 1

17. Primary Outcome: Number of Infants With a Child Behavior Checklist for Ages 1.5 to 5 Years (CBCL/1.5 to 5) Score Above the 97th Percentile for a Subset of Prespecified Questions That Relate to Attention and Hyperactivity Problems
Description: The CBCL/1.5 to 5 questionnaire is a parent-completed questionnaire used for assessing behavioral problems and social competencies. It included approximately 100 items that described specific kinds of behavioral, emotional, and social problems that characterized preschool children between the ages of 1.5 and 5 years. Each question could be answered as "not true scored as"0",somewhat or sometimes true scored as"1"or very true or often true scored as "2". There were 6 questions related to attention and hyperactivity problems. The responses to those 6 questions were summed (ranged 0 to 12). Total score of 0 to 9 indicated normal, 10 indicated borderline and 11 to 12 indicated significant attention and hyperactivity problems. Scores above the 97th percentile are in the significant range of clinical concern. Number of infants with CBCL/1.5 to 5 score above 97th percentile for subset of pre-specified questions related to attention and hyperactivity problems at 24 months is reported.
Time Frame: At 24 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 2 | 12 | 14
Participants | 0 | 1 | 0

18. Primary Outcome: Number of Infants Indicated as Needing Further Evaluation After Completion of the Modified Checklist for Autism in Toddlers- Revised With Follow-up (M-CHAT-R/F)
Description: The M-CHAT-R/F is a parent-reported autism screening tool designed to identify children 16 to 30 months of age who received a more thorough assessment for possible early signs of autism spectrum disorder (ASD) or developmental delay. The M-CHAT-R/F consisted of 20 questions that were answered with either "yes, scored as 0" or "no, scored as 1". Total scores (ranged 0 to 20) on the M-CHAT-R/F between 0 and 2 indicated a low risk, scores between 3 and 7 indicated a medium risk and triggered administration of the follow-up questionnaire, and scores between 8 and 20 indicated a high risk. Number of infants who needed further evaluation as per the M-CHAT-R/F at 18 and 24 months is presented.
Time Frame: 18 and 24 months
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 2 | 11 | 13
Participants
  18 months,n=2,10,7: number analyzed (Participants) | 2 | 10 | 7
  18 months,n=2,10,7 | 0 | 0 | 0
  24 months,n=2,11,13 | 0 | 0 | 0

19. Primary Outcome: Number of Infants Referred for Neurological Evaluation to Determine Diagnosis of Cerebral Palsy
Description: Parents reported in CHI questionnaire if their infant had cerebral palsy. If the infant was not diagnosed with cerebral palsy, then this was detected as part of the ASQ-3 assessment, based on the results of the gross motor scale. To confirm the diagnosis of cerebral palsy, the healthcare practitioner referred the infant for further neurological tests if they scored in the black zone of the ASQ-3 at the month 24 assessment. Number of infants referred for neurological evaluation to determine diagnosis of cerebral palsy at 24 months is presented.
Time Frame: At 24 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 2 | 19 | 25
Participants | 0 | 0 | 0

20. Primary Outcome: Number of Infants With the Indicators of Neurodevelopmental Impairment
Description: The indicators of neurodevelopmental impairment were 'hearing impaired, uncorrected even with aids'; 'blindness in 1 or both eyes, or sees light only'; 'cerebral palsy-moderate and severe (moderate: Grade 2 or 3 using the gross motor functional classification system [GMFCS] and severe: Grade 4 or 5 using the GMFCS)'; 'cognitive impairment: BSID-III cognitive scale score of less than 2 SDs below mean score (less than 4)'; 'motor impairment: BSID-III motor composite scale score of greater than 2 SDs below mean score (less than 70)'; 'diagnosis of ASD, attention deficit disorder (ADD) or attention deficit hyperactivity disorder (ADHD)'. Number of infants having any 1 of these indicators is presented.
Time Frame: Up to 24 months
Population: ARIOS Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
Number analyzed (Participants) | 4 | 30 | 36
Participants
  Hearing impaired, uncorrected even with aids | 0 | 0 | 0
  Blindness in 1 or both eyes, or sees light only | 0 | 0 | 0
  Cerebral palsy (moderate and severe) | 0 | 0 | 0
  Cognitive impairment | 0 | 1 | 1
  Motor impairment | 0 | 1 | 1
  Diagnosis of ASD,ADD or ADHD | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) were collected for infants from after 28 days post estimated due date until maximum of 24 months chronological age. Non-SAEs were not collected, since all the adverse events that occurred in infants were considered as SAEs
Description: SAEs were reported for ARIOS Safety Population which comprised of a subset of Infant Safety Population (all the infants whose mothers were randomized and received retosiban or comparator in any of the Phase III treatment trials) for which the mother/infant pairs were enrolled into the ARIOS study.
Arm/Group | Placebo (200719 Study) | Atosiban (200721 Study) | Retosiban (200719 and 200721 Study)
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/44 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/5 | 6/44 | 3/49
Other Adverse Events (participants affected / at risk) | 0/5 | 0/44 | 0/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (200719 Study) (N=5) | Atosiban (200721 Study) (N=44) | Retosiban (200719 and 200721 Study) (N=49)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Acute bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (4)
Congenital cataract (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Injury of genitals (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Congenital hydrocoele (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumococcal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Acute pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Cervical lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Circumoral cyanosis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-01): https://cdn.clinicaltrials.gov/large-docs/84/NCT02292784/Prot_000.pdf
  • Statistical Analysis Plan (2019-12-05): https://cdn.clinicaltrials.gov/large-docs/84/NCT02292784/SAP_001.pdf